CLINICAL TRIAL: NCT02316899
Title: Phase III Study of ASP0456 - A Double-blind, Placebo-controlled, Parallel-group, Comparative Study and Long-term Study in Patients With Irritable Bowel Syndrome With Constipation (IBS-C)
Brief Title: Phase III Study to Evaluate the Efficacy and Safety of ASP0456 in Patients With Constipation Predominant Irritable Bowel Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0456-CL-0031
Record Dates: First submitted 2014-12-04; First posted 2014-12-15 (Estimated); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Irritable Bowel Syndrome With Constipation (IBS-C)
Keywords: ASP0456; constipation; linaclotide; irritable bowel syndrome (IBS)
MeSH Terms: conditions — Constipation; Irritable Bowel Syndrome | interventions — linaclotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ASP0456 (Period I) (Experimental): Up to 12 weeks
  Interventions: Drug: linaclotide
- Placebo (Period I) (Placebo Comparator): Up to 12 weeks
  Interventions: Drug: Placebo
- ASP0456 (Period II) (Experimental): From 12 weeks to 52 weeks
  Interventions: Drug: linaclotide

INTERVENTIONS:
Drug: linaclotide — Oral administration once daily
  Other Names: ASP0456
  Arms: ASP0456 (Period I); ASP0456 (Period II)
Drug: Placebo — Oral administration once daily
  Arms: Placebo (Period I)

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of ASP0456 in patients with constipation predominant irritable bowel syndrome (IBS-C).

DETAILED DESCRIPTION:
<Period I (double-blind period)> A multicenter, collaborative, double-blind, parallel comparative study is conducted using IBS-C patients as subjects to verify efficacy of ASP0456 and examine the safety. After the 2-week bowel habit observation period, subjects satisfying the primary enrollment criteria are randomly allocated to either ASP0456 group or placebo group, and orally administered the drug or placebo once daily before breakfast for 12 weeks.

<Period II (non-blind period)> A multicenter, collaborative, non-blind, non-controlled study is conducted to examine safety and efficacy of ASP0456 in long-term administration in IBS-C patients. After Period I, subjects satisfying the transfer criteria are orally administered ASP0456 once daily before breakfast for 40 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had abdominal pain or discomfort repeatedly for at least 3 days per month during the 3 months before screening examination associated with at least 2 out of the following 3 conditions: (1) Improvement with defecation; (2) Onset associated with a change in frequency of stool; and (3) Onset associated with a change in form (appearance) of stool, and had the above symptom (IBS symptom) 6 months or more before the screening examination period
* Patients with ≥ 25% of stools hard or lumpy (with each bowel movement occurring without antidiarrheal, laxative, suppository or enema) and <25% of them loose (mushy) or watery during the 3 months before the screening examination
* Patients who had pancolonoscopy or contrast enema (or sigmoidoscopy) after the onset of IBS symptom and had no organic changes

Exclusion Criteria:

* Patient with history of surgical resection of stomach, gallbladder, small intestine, or large intestine (excluding resection of appendicitis and benign polyp)
* Patient with history or current affection of inflammatory bowel disease (Crohn's disease or ulcerative colitis)
* Patient with history or current affection of ischemic colitis
* Patient currently affected by infectious enteritis
* Patient currently affected by hyperthyroidism or hypothyroidism
* Patient currently affected by active peptic ulcer
* In the case of a female patient, the one currently affected by endometriosis or uterine adenomyosis
* Patient with high depression or anxiety considered to influence drug evaluation
* Patient with history of abuse of drug or alcohol within a year before consent acquisition, or with current abuse
* Patient who used or underwent or will use or undergo drug/therapy/test prohibited to combine 3 days before the start of bowel habit observation period (Day -17) or thereafter
* Patient with history or current affection of malignant tumor
* Patient currently affected by serious cardiovascular disease, respiratory disease, kidney disease, hepatic disease, gastrointestinal disease (excluding IBS), hemorrhagic disease, or neural/mental disease
* Patient with history of drug allergy

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2014-10-21 (Actual); Primary Completion 2015-09-19 (Actual); Study Completion 2016-03-29 (Actual)

PRIMARY OUTCOMES:
Responder rate of Global assessment of relief of IBS symptoms during 12 weeks. | During 12 weeks
  The responder of the evaluation items during the 12 weeks shall be the subject satisfying weekly responder of the evaluation items for over 6 weeks of the 12 weeks.
Responder rate of CSBM during 12 weeks | During 12 weeks
  CSBM: Complete Spontaneous Bowel Movement. The responder of the evaluation items during the 12 weeks shall be the subject satisfying weekly responder of the evaluation items for over 6 weeks of the 12 weeks.

SECONDARY OUTCOMES:
Responder rate of SBM during 12 weeks | During 12 weeks
  SBM: Spontaneous Bowel Movement
Responder rate of Abnormal bowel habits improvement during 12 weeks | During 12 weeks
Responder rate of Abdominal pain/discomfort relief during 12 weeks | During 12 weeks
Weekly responder rate of Global assessment of relief of IBS symptoms | Up to 52 weeks
  The weekly responder of the evaluation items shall be the subject satisfying the followings at the time of evaluation in each week.Score of Global assessment of relief of IBS symptoms (7 scores: 1-7) is 1 or 2
Weekly responder rate of CSBM | Up to 52 weeks
  Weekly responder of CSBM: The weekly mean value of CSBM frequency is more than 3 and over 1 more than the weekly mean value of CSBM frequency in the bowel habit observation period
Weekly responder rate of SBM | Up to 52 weeks
  Weekly responder of SBM: The weekly mean value of SBM frequency is more than 3 and over 1 more than the weekly mean value of SBM frequency in the bowel habit observation period
Weekly responder rate of Abnormal bowel habits improvement | Up to 52 weeks
  Score of abdominal bowel habits improvement effect (7 scores: 1-7) is 1 or 2
Weekly responder rate of Abdominal pain/discomfort relief | Up to 52 weeks
  Score of abdominal pain/discomfort improvement effect (7 scores: 1-7) is 1 or 2.
Changes in weekly average of SBM frequency, CSBM frequency, stool form scores, abdominal pain/discomfort severity, abdominal bloating severity, and straining severity. | From baseline to every week until 52 weeks
Changes in IBS-QOL-J scores (entire scores or scores on the sub-scales) | Weeks 0, 4, 8, 12, 16, 20, 24, 28, 40, 52
  IBS-QOL-J: Irritable bowel syndrome quality of life Japanese version
Percentage of subjects with SBM within 24 hours after start of the initial administration | Up to 24 hours
Percentage of subjects with CSBM within 24 hours after start of the initial administration | Up to 24 hours
Safety assessed by development of incidence of adverse events, vital signs, and clinical laboratory tests | Up to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (61):
- Japan (61):
  - Site JP00004, Aichi
  - Site JP00048, Aichi
  - Site JP00049, Aichi
  - Site JP00038, Chiba
  - Site JP00039, Chiba
  - Site JP00040, Chiba
  - Site JP00041, Chiba
  - Site JP00042, Chiba
  - Site JP00002, Fukuoka
  - Site JP00060, Fukuoka
  - Site JP00061, Fukuoka
  - Site JP00001, Hokkaido
  - Site JP00006, Hokkaido
  - Site JP00007, Hokkaido
  - Site JP00057, Hyōgo
  - Site JP00058, Hyōgo
  - Site JP00059, Hyōgo
  - Site JP00030, Kanagawa
  - Site JP00031, Kanagawa
  - Site JP00032, Kanagawa
  - Site JP00033, Kanagawa
  - Site JP00034, Kanagawa
  - Site JP00035, Kanagawa
  - Site JP00036, Kanagawa
  - Site JP00037, Kanagawa
  - Site JP00056, Kyoto
  - Site JP00003, Osaka
  - Site JP00050, Osaka
  - Site JP00051, Osaka
  - Site JP00052, Osaka
  - Site JP00053, Osaka
  - Site JP00054, Osaka
  - Site JP00055, Osaka
  - Site JP00043, Saitama
  - Site JP00044, Saitama
  - Site JP00045, Saitama
  - Site JP00046, Saitama
  - Site JP00047, Saitama
  - Site JP00005, Tokyo
  - Site JP00008, Tokyo
  - Site JP00009, Tokyo
  - Site JP00010, Tokyo
  - Site JP00011, Tokyo
  - Site JP00012, Tokyo
  - Site JP00013, Tokyo
  - Site JP00014, Tokyo
  - Site JP00015, Tokyo
  - Site JP00016, Tokyo
  - Site JP00017, Tokyo
  - Site JP00018, Tokyo
  - Site JP00019, Tokyo
  - Site JP00020, Tokyo
  - Site JP00021, Tokyo
  - Site JP00022, Tokyo
  - Site JP00023, Tokyo
  - Site JP00024, Tokyo
  - Site JP00025, Tokyo
  - Site JP00026, Tokyo
  - Site JP00027, Tokyo
  - Site JP00028, Tokyo
  - Site JP00029, Tokyo

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Fukudo S, Miwa H, Nakajima A, Haruma K, Kosako M, Nakagawa A, Akiho H, Yamaguchi Y, Johnston JM, Currie M, Kinoshita Y. A randomized controlled and long-term linaclotide study of irritable bowel syndrome with constipation patients in Japan. Neurogastroenterol Motil. 2018 Dec;30(12):e13444. doi: 10.1111/nmo.13444. Epub 2018 Aug 22. PMID 30136447
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=207